CLINICAL TRIAL: NCT01512121
Title: Investigating the Cortical Correlates of Spinal Cord Stimulation Using Functional Magnetic Resonance Imaging
Brief Title: Spinal Cord Stimulation and Functional MRI
Status: Completed | Type: Observational
Sponsor: Vibhor Krishna (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Vibhor Krishna, Assistant Professor of Neurological Surgery, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2011H0040
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Complex Regional Pain Syndrome (CRPS); Neuropathic Leg Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- functional MRI testing: fMRI scanning with SCS "on" and "off" at different settings.

SUMMARY:
The overall objective of this study is to assess patterns of fMRI cortical activation with spinal cord stimulation (SCS) in patients with neuropathic leg pain and therefore define cortical correlates, as well as to investigate cortical representations of pain and pain relief and the interactions therein, in the setting of neuropathic leg pain and SCS.

DETAILED DESCRIPTION:
The main objective is to define, using functional magnetic resonance imaging, the effects of spinal cord stimulation (SCS) on cortical and subcortical BOLD effects in patients with neuropathic leg pain. Our hypothesis is that SCS will demonstrate a consistent pattern of BOLD activation that will correlate with symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years at time of enrollment.
* Have previous implantation of thoracic epidural Medtronic Restore Ultra, Prime Advanced and Restore Advanced SCS in place for the treatment of CPRS-type 1 or chronic refractory neuropathic leg pain following FBSS. The implantation must be 3 or more months prior to enrollment.
* Patient must have reported significant pain improvement (>50%) following implantation of the SCS.
* Have consistently reproducible pain relief (> 50%) within 10 minutes of switching SCS from an OFF state to an ON state (with "optimal" parameters - see below).
* The SCS battery is implanted in the buttocks region.
* Unilateral or bilateral extremity pain.
* Able to provide informed consent.

Exclusion Criteria:

- Contraindication to MRI such as: SCS lead in the cervical epidural region Cardiac pacemaker Intracranial aneurysm clips, metallic implants or external clips within 10mm of the head Metallic foreign metals within the orbits Pregnancy; (urine pregnancy test will be done to confirm) Claustrophobia

* Pattern of response to spinal cord stimulation Inconsistent response of pain to spinal cord stimulation Long interval (> 10 minutes) before pain relief following switching SCS from an OFF state to an ON state (with "optimal" parameters) - long "washout" period Lack of significant pain improvement (< 50%) following implantation of SCS
* Positive history of significant brain lesions or pathology including:
* Prior ablative neurosurgery
* History of large vessel strokes or brain tumors
* Psychological Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with implanted spinal cord stimulators
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Effects of spinal cord stimulation on patients with neuropathic leg pain through fMRI analysis | 1 year
  We are analyzing the data from fMRI scans to understand more the functional activation of the cerebral cortex

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor Krishna, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Medical Center, Columbus, Ohio, United States